CLINICAL TRIAL: NCT01624727
Title: Slowing HEART diSease With Lifestyle and Omega-3 Fatty Acids (HEARTS)
Brief Title: Slowing HEART diSease With Lifestyle and Omega-3 Fatty Acids
Acronym: HEARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Tufts Medical Center (Other)
Responsible Party: Principal Investigator, Francine K. Welty, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006P000175; P50HL083813 (NIH)
Record Dates: First submitted 2012-05-15; First posted 2012-06-21 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Coronary Heart Disease; Metabolic Syndrome
Keywords: Coronary heart disease; metabolic syndrome; CT angiography
MeSH Terms: conditions — Coronary Disease; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Those randomized to usual care will continue to follow the care provided by their cardiologist. They will have all the follow-up phone calls, visits and testing which the intervention group has.
- Lovaza (Omega 3 ethyl esters) (Active Comparator)
  Interventions: Dietary Supplement: Omega 3 acid ethyl esters

INTERVENTIONS:
Dietary Supplement: Omega 3 acid ethyl esters — Lovaza 3.6 g daily
  Arms: Lovaza (Omega 3 ethyl esters)

SUMMARY:
The purpose of the study is to target inflammation to reduce progression of noncalcified plaque in the coronary arteries using omega-3 fatty acid supplementation compared to standard of care.

DETAILED DESCRIPTION:
Study Design: This is a randomized, parallel study design with a usual care control group. 278 subjects with coronary heart disease (CHD) are being randomized to omega-3 supplementation or standard of care (139 in each arm).

Multidetector computed tomographic angiography (MDCTA) is performed at baseline to quantitate the amount of noncalcified and calcified coronary plaque and again at 30 month follow-up to determine if there has been a change in the volume of noncalcified or total plaque. The primary endpoint is change in coronary noncalcified plaque volume during the 30 months of intervention between active and standard of care.

Hypothesis: Percent change in progression of coronary plaque volume will be less for the omega-3 fatty acid intervention compared to standard of care.

Secondary endpoints include plasma levels of inflammatory markers, lipids and measures of insulin sensitivity.

Secondary outcomes include testing the hypothesis that targeting inflammation with omega-3 fatty acids will be associated with:

1. Change in total plaque volume per patient.
2. improvement in physical function and exercise and reduction in pain and stiffness as measured by the WOMAC questionnaire
3. Reduction of mediators of inflammation in the circulation including CRP, PAI-1, serum amyloid A, MMP-9 and fibrinogen, pro-inflammatory cytokines including IL-6, TNF-a and IL-1b, the adhesion molecules VCAM-1 and ICAM-1, increase in adiponectin and reduction in serum nitrotyrosine as a marker of oxidative stress.
4. Reduction of insulin resistance assessed by fasting insulin and homeostasis model assessment of insulin resistance (HOMA-IR).
5. Reduction of inflammation in the liver associated with nonalcoholic steatohepatitis (NASH), a newly recognized component of the metabolic syndrome, and reduction of fatty liver quantitated by computerized tomography and levels of AST and ALT as markers of liver inflammation related to NASH.
6. Investigation of the relationship between vitamin D status and coronary plaque progression as well as with insulin resistance (HOMA-IR), beta-cell function (HOMA-%beta) and inflammatory cytokines.
7. Determination of whether baseline vitamin D levels predict clinical response to the omega-3 fatty acid intervention, and whether hypovitaminosis D is associated with plaque progression.

ELIGIBILITY:
Inclusion Criteria:

1. coronary artery disease
2. previous myocardial infarction
3. angioplasty (> 6 months ago)
4. previous coronary bypass surgery (> 12 months ago)
5. stable angina
6. non-calcified plaque on prior CT
7. abnormal exercise tolerance test
8. aged 21- 80 years
9. BMI ≥ 27 kg/m2 and ≤ 35 kg/m2 if female and ≤ 40 kg/m2 if male (a BMI > 24.5 for subjects from Asian origin)
10. stable dose of statin for 1 month at screening or unable to tolerate a statin
11. normal renal function - estimated creatinine clearance calculated using Cockcroft-Gault (CG) equation ≥60 at screening [eCrCLCG (ml/min) = [(140 - age) x weight (kg)]/[SCr(mg/dl) x 72] x [0.85 if female] or serum Cr < 1.3
12. ALT, AST) < 3 times upper limits of normal)
13. normal thyroid function or on stable dose replacement therapy
14. an ETT performed within 12 months prior

Exclusion criteria

1. unstable angina (increase in frequency or severity of anginal episodes or development of chest pain at rest)
2. significant obstructive disease in left main coronary artery, ostial LAD or newly diagnosed three-vessel disease since prior cardiac catheterization by MDCTA
3. significant heart failure (NYHA class III and IV)
4. Current atrial fibrillation or Wolf-Parkinson-White (WPW) syndrome
5. allergy to beta-blocker in subjects with resting heart rate > 65 bpm
6. systolic blood pressure > 160 mm Hg
7. diastolic BP > 100 mm Hg
8. persons with allergies to iodinated contrast material or shellfish
9. allergy to nitroglycerin
10. history of asthma only if unable to tolerate beta-blockers
11. BMI > 35 kg/m2 if female and > 40 kg/m2 if male
12. body weight > 350 lbs
13. Use of drugs for weight loss [eg Xenical (orlistat), Meridia (sibutramine), Acutrim (phenylpropanolamine) or similar over-the-counter medications] within three months of screening
14. surgery within 30 days of screening
15. history of acquired immune deficiency syndrome or human immunodeficiency virus (HIV)
16. poor mental function or history of dementia/Alzheimer's Disease or on medications used for treatment of dementia [e.g. Tacrine (Cognex), Rivastigmine (Exelon), Galantamine (Razadyne, Reminyl), Donepezil (Aricept), Memantine (Namenda)] or any other reason to except patient difficulty in complying with the requirements of the study
17. medicine for erectile dysfunction within 72 hours prior to MDCTA
18. Prior stroke with residual cognitive deficit or functional deficit preventing any type of exercise
19. Current chemotherapy or radiation for malignancy
20. Current weekly alcohol consumption > 21 units/week (1 unit = 1 beer, 1 glass of wine, 1 mixed cocktail containing 1 ounce of alcohol)

Exclusions based on nuclear imaging:

1. Transient cavity dilation
2. More than one vascular territory involved with reversible defect (multiple defects)
3. Reversible defects involving the anterior wall, septum or apex (LAD territory)

Exclusions based on echocardiography imaging:

1. More than one vascular territory involved with inducible wall motion abnormalities (multiple defects) 2. Inducible wall motion abnormalities involving the anterior wall, septum or apex (LAD territory)

-

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2009-06; Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is change in coronary noncalcified plaque volume. | Baseline and 30 months
  MDCTA is performed at baseline to quantitate the amount of noncalcified and calcified coronary plaque and again at 30 month follow-up to determine if there has been a change in the volume of noncalcified or total plaque. The primary endpoint is change in coronary noncalcified plaque volume during the 30 months of intervention between active and standard of care. The hypothesis is that those on Lovaza will have less progression of coronary plaque compared to those in usual care.

SECONDARY OUTCOMES:
Coronary artery plaque assessment | Baseline and 30 months
  1. Percent atheroma volume calculated as the proportion of the entire vessel wall occupied by atherosclerotic plaque and total atheroma volume, normalized to segment length.
  2. Maximum percent diameter stenosis and minimal luminal diameter.
  3. Number of subjects with categorical variables of maximal stenosis >50% and number with 3-vessel disease >20%.
  4. Number of subjects with stenosis of 0-29%, 30-49%, 50-69% and >70% stenosis at baseline compared to 30 months.
  5. Change in remodeling index - ratio of plaque volume at the most diseased site compared to the least diseased site.
Effect of Lovaza on Physical Function, Pain, Stiffness and Exercise | Baseline and 1 year
  Those on Lovaza will have better physical function and less pain and stiffness as assessed by the WOMAC questionnaire and more minutes of exercise per week compared to control
Inflammatory markers | Baseline and 30 months
  Compared to usual care, those on Lovaza will have reduction of mediators of inflammation in the circulation, including CRP, PAI-1, serum amyloid A, MMP-9 and fibrinogen, pro-inflammatory cytokines including IL-6, TNF-a and IL-1b, the adhesion molecules VCAM-1 and ICAM-1, increase in adiponectin and reduction in serum nitrotyrosine as a marker of oxidative stress. Additional inflammatory markers may be identified in the future and measured.
Pericardial Fat | Baseline and 30 months
  The amount of pericardial fat will be quantitated by CT at baseline and 30-month follow-up. The percent change between the two time-frames will be measured. Those on Lovaza and/or those who have lost weight will have a reduction (or lack of increase) in pericardial fat at 30-months compared to those in usual care.
Insulin Resistance | Baseline and 30 months
  Insulin resistance will be assessed by fasting insulin and homeostasis model assessment of insulin resistance (HOMA-IR) at baseline and 30-months in the two study groups.
Nonalcoholic steatohepatitis (NASH) | Baseline and 30 months
  Reduction of inflammation in the liver associated with nonalcoholic steatohepatitis (NASH), a component of the metabolic syndrome, and reduction of fatty liver quantitated by computerized tomography and levels of AST and ALT as markers of liver inflammation related to NASH.
Vitamin D Levels and coronary plaque progression | Baseline and 30 months
  1. Investigation of the relationship between vitamin D status and coronary plaque progression, insulin resistance (HOMA-IR), beta-cell function (HOMA-%beta) and inflammatory cytokines
  2. Do baseline vitamin D levels predict response to omega-3 fatty acid supplementation?
Cognitive function | Baseline, 1 year and 30-months
  To determine if those on Lovaza have less decline in cognitive function at 1 year and 30 months of follow-up compared to those in the usual care group.
Exercise capacity and coronary plaque | Baseline
  To determine if exercise capacity correlates with coronary plaque measurements. The hypothesis is that those with better exercise capacity will have lower amounts of coronary plaque.
Urinary microalbumin and coronary plaque | Baseline and 30-months
  At baseline, subjects with lower urinary microalbumin will have lower amounts of coronary plaque. Those taking Lovaza will have less increase in urinary microalbmumin at 30-month follow-up compared to those in usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Francine K Welty, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - South Shore Medical Group, Milton, Massachusetts

REFERENCES:
- [Derived] Ahmad B, Daher R, Malik A, Jeong YN, Welty FK. Omega-3 fatty acids and oral and systemic inflammation: A secondary analysis of a randomized trial in patients with coronary artery disease. J Am Dent Assoc. 2026 Feb 5:S0002-8177(25)00757-3. doi: 10.1016/j.adaj.2025.12.013. Online ahead of print. PMID 41642164
- [Derived] Welty FK, Hariri E, Asbeutah AA, Daher R, Amangurbanova M, Chedid G, Elajami TK, Alfaddagh A, Malik A. Regression of Coronary Fatty Plaque and Risk of Cardiac Events According to Blood Pressure Status: Data From a Randomized Trial of Eicosapentaenoic Acid and Docosahexaenoic Acid in Patients With Coronary Artery Disease. J Am Heart Assoc. 2023 Sep 19;12(18):e030071. doi: 10.1161/JAHA.123.030071. Epub 2023 Sep 8. PMID 37681568
- [Derived] Chedid G, Malik A, Daher R, Welty FK. Higher exercise capacity, but not omega-3 fatty acid consumption, predicts lower coronary artery calcium scores in women and men with coronary artery disease. Atherosclerosis. 2023 Nov;384:117168. doi: 10.1016/j.atherosclerosis.2023.06.074. Epub 2023 Jun 26. PMID 37541921
- [Derived] Welty FK, Schulte F, Alfaddagh A, Elajami TK, Bistrian BR, Hardt M. Regression of human coronary artery plaque is associated with a high ratio of (18-hydroxy-eicosapentaenoic acid + resolvin E1) to leukotriene B4. FASEB J. 2021 Apr;35(4):e21448. doi: 10.1096/fj.202002471R. PMID 33749913
- [Derived] Malik A, Ramadan A, Vemuri B, Siddiq W, Amangurbanova M, Ali A, Welty FK. omega-3 Ethyl ester results in better cognitive function at 12 and 30 months than control in cognitively healthy subjects with coronary artery disease: a secondary analysis of a randomized clinical trial. Am J Clin Nutr. 2021 May 8;113(5):1168-1176. doi: 10.1093/ajcn/nqaa420. PMID 33675344
- [Derived] Malik A, Kanduri JS, Asbeutah AAA, Khraishah H, Shen C, Welty FK. Exercise Capacity, Coronary Artery Fatty Plaque, Coronary Calcium Score, and Cardiovascular Events in Subjects With Stable Coronary Artery Disease. J Am Heart Assoc. 2020 Apr 7;9(7):e014919. doi: 10.1161/JAHA.119.014919. Epub 2020 Mar 26. PMID 32212910
- [Derived] Alfaddagh A, Elajami TK, Saleh M, Mohebali D, Bistrian BR, Welty FK. An omega-3 fatty acid plasma index >/=4% prevents progression of coronary artery plaque in patients with coronary artery disease on statin treatment. Atherosclerosis. 2019 Jun;285:153-162. doi: 10.1016/j.atherosclerosis.2019.04.213. Epub 2019 Apr 13. PMID 31055222
- [Derived] Alfaddagh A, Elajami TK, Ashfaque H, Saleh M, Bistrian BR, Welty FK. Effect of Eicosapentaenoic and Docosahexaenoic Acids Added to Statin Therapy on Coronary Artery Plaque in Patients With Coronary Artery Disease: A Randomized Clinical Trial. J Am Heart Assoc. 2017 Dec 15;6(12):e006981. doi: 10.1161/JAHA.117.006981. PMID 29246960
- [Derived] Elajami TK, Alfaddagh A, Lakshminarayan D, Soliman M, Chandnani M, Welty FK. Eicosapentaenoic and Docosahexaenoic Acids Attenuate Progression of Albuminuria in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease. J Am Heart Assoc. 2017 Jul 14;6(7):e004740. doi: 10.1161/JAHA.116.004740. PMID 28710178